CLINICAL TRIAL: NCT00552006
Title: A Randomized Controlled Clinical Trial (RCCT) to Test the Effectiveness of Narrative Exposure Therapy (NET) Versus an Attention Control Condition (AC) in Reducing Trauma Related Symptoms in Formerly Abducted Children and Former Child Soldiers Suffering From Posttraumatic Stress Disorder (PTSD)
Brief Title: Treatment of Formerly Abducted Children (FAC) in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Prof.Dr. Frank Neuner, Bielefeld University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE 1390/2-1
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2008-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Treatment; Randomized Controlled Clinical Trial; Combat; Child Soldiers; Dissemination; Narrative Exposure Therapy; Africa
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NET (Experimental)
  Interventions: Behavioral: Narrative Exposure Therapy
- AC (Active Comparator)
  Interventions: Behavioral: Academic Counseling
- WL (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Narrative Exposure Therapy (NET) is based on Testimony Therapy in combination with cognitive behavioural exposure techniques and elements of client-centered counselling. In cooperation with the therapist the clients can restore their autobiographic memories about their traumatic experiences. In this way fragmentary memories are transformed into a coherent narrative structure. This practice enables the processing of painful emotions and the construction of clear contingencies of dangerous and safe conditions, generally leading to significant emotional recovery. Therapeutic aims are the reduction of PTSD-Symptomload via activation of fear-network and habituation of fear and the placement of traumatic experiences in a reconstructed, detailed and consistent autobiography.
  NET will be applied in eight sessions (90-120min/session) in a standardized, manualized manner.
  Other Names: NET
  Arms: NET
Behavioral: Academic Counseling — Missing time in educational life is one major issue for formerly abducted people. The Academic Counseling (AC) intervention is an active Control condition and improves English skills and works at the same time on concentration, learning and memory abilities. The clients will gain some of the abilities and skills they might have lost or developed weaknesses in due to their abduction.
  AC will be applied in eight sessions (90-120min/session) in a standardized, manualized manner.
  Other Names: AC
  Arms: AC

SUMMARY:
In the aftermath of traumatic experiences like natural disasters or man-caused traumatic events, such as war experiences, a substantial part of the affected individuals develop a number of psychological symptoms. The characteristic symptom pattern occurring in the aftermath of traumatic events is called posttraumatic stress disorder (PTSD) and includes functional impairment of the affected individuals. The investigators want to test whether Narrative Exposure Therapy (NET) is an effective tool in reducing trauma related symptoms in formerly abducted children and youths and former child soldiers, when applied by lay personnel.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of PTSD (Post-Traumatic Stress Disorder) derived from expert interviews
* member of the group of formerly abducted people or former child soldiers

Exclusion Criteria:

* current substance dependence
* mental retardation
* psychotic disorder

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Load of traumatic symptoms measured via the CAPS (Clinician-administered PTSD scale) | 3 months, 6 months and 1 year after completion of treatment

SECONDARY OUTCOMES:
Load of depressive symptoms measured via the MINI, strength of suicidal ideation measured via the MINI, functionality measured via the CAPS, feelings of guilt measured via the CAPS, stigmatization measured via an adapted version of the PSQ | 3 months, 6 months and 1 year after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank Neuner, Univ.-Prof. Dr., Principal Investigator — Bielefeld University; Thomas Elbert, Univ.-Prof. Dr., Principal Investigator — University of Konstanz; Verena Ertl, Dipl.-Psych. (MSc), Study Director — Bielefeld University
Locations (1):
- Vivo Counselling Centre, Anaka, Amuru, Uganda

REFERENCES:
- [Derived] Ertl V, Pfeiffer A, Schauer E, Elbert T, Neuner F. Community-implemented trauma therapy for former child soldiers in Northern Uganda: a randomized controlled trial. JAMA. 2011 Aug 3;306(5):503-12. doi: 10.1001/jama.2011.1060. PMID 21813428